CLINICAL TRIAL: NCT05548088
Title: An Exploratory Clinical Study of the Safety and Efficacy of LILRB4 STAR-T Cells for the Treatment of Relapsed/Refractory Acute Myeloid Leukemia/Chronic Granulocytic-Mononocytic Leukemia
Brief Title: LILRB4 STAR-T Cells in the Treatment of R/R AML/CMML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Bristar Immunotech Limited (Unknown)
Responsible Party: Principal Investigator, Xiangyu Zhao, associate professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YTS104-002
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia and Chronic Granulocytic-Mononocytic Leukemia
Keywords: LILRB4 STAR-T cells
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LILRB4 STAR-T cells (Experimental): The subjects met the inclusion criteria, then collect the Lymphocytes and transfected with lentivirus to obtain LILRB4 STAR-T cells. The subjects were given fludarabine and cyclophosphamide chemotherapy 5 days before and 3 days after cell reinfusion. After two days of rest, the cells were reinjected at doses of 1E6,3E6,6E6,and 1E7/kg.
  Interventions: Biological: LILRB4 STAR-T cells

INTERVENTIONS:
Biological: LILRB4 STAR-T cells — Subjects with relapsed/refractory acute myeloid leukemia will be enrolled in the study, and Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4and-3followed by infusion of STAR-T cells. STAR-T cells will be intravenously infused with a escalated dose of 1E6,3E6,6E6,1E7 cells/kg

SUMMARY:
This study is an exploratory study to evaluate the safety, tolerability, and efficacy of LILRB4 STAR-T cells in relapsed and refractory acute myeloid leukemia/Chronic Granulocytic-Mononocytic Leukemia subjects.

DETAILED DESCRIPTION:
This study will recruit LILRB4 positive AML/Chronic Granulocytic-Mononocytic Leukemia subjects,and Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of LILRB4 STAR-T cells. LILRB4 STAR-T cells will be intravenously infused with a escalated dose of 1E6, 3E6, 6E6, 1E7 cells/kg.Safety and efficacy of LILRB4 STAR-T cells therapy will be monitored.The primary endpoint of the study is to observe DLT, AE, SAE, CRS and ICANS. Secondary objectives are to observe the efficacy of LILRB4 STAR-T cells, including Disease response, CR rate, ORR, RFS, EFS, OS, PK, PD and ADA.

ELIGIBILITY:
Inclusion Criteria:

(A) Subjects must meet all of the following enrollment criteria to be enrolled in this study.

1. Age ≥ 18 years,≤ 60 years and gender;
2. Patients with acute myeloid leukemia or chronic granulomonocytic leukemia; 1) Patients with acute myeloid leukemia (AML) diagnosed according to the World Health Organization (WHO) 2016 criteria and who should meet any of the following relapsed-refractory (R/R) AML according to the Chinese Guidelines for the Diagnosis and Treatment of Relapsed-Refractory Acute Myeloid Leukemia (2021 Edition):

   * Primary patients who have failed 2 courses of treatment with a standard regimen (containing cytarabine and an anthracycline or anthraquinone);
   * Those who relapsed within 12 months after complete remission (CR) with consolidation and intensive therapy;
   * Those who relapsed after 12 months but failed to respond to conventional treatment;
   * Those with 2 or more recurrences;
   * Those with persistent extramedullary leukemia. Note: Definition of relapse: reappearance of leukemic cells in the peripheral blood or >5% of primitive cells in the bone marrow after CR (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extraparenchymal infiltration of leukemic cells.

     2) Chronic granulocytic-monocytic leukemia diagnosed according to the World Health Organization (WHO) 2016 Classification Criteria for Tumors of Hematopoietic and Lymphoid Tissues and the Chinese Guidelines for the Diagnosis and Treatment of Chronic Granulocytic-Mononocytic Leukemia (2021 edition), with relapse refractory defined as follows: at least 2 complete cycles of at least one treatment (e.g., demethylating drugs ) or allogeneic hematopoietic stem cell transplantation (allo-HSCT) ) without achieving remission or relapse after remission.
3. ECOG score 0-2;
4. Bone marrow samples were positive for LILRB4 (flow-through assay);
5. Good organ function:

   Liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN), alanine transaminase (AST), alanine transaminase (ALT) ≤ 3 x ULN; Renal function: serum creatinine (Cr) ≤ 1.5 x ULN or creatinine clearance (Cockcroft-Gault formula) ≥ 60 mL/min; Cardiac function: left ventricular ejection fraction (LVEF) ≥50%; Pulmonary function: defined as ≤ grade 1 dyspnea and oxygen saturation > 92%.
6. Female subjects of childbearing age or male subjects whose partner is a woman of childbearing age agree to use an effective method of contraception throughout the trial and for 12 months after cell infusion;
7. Subjects voluntarily enrolled in the study, signed an informed consent form, were compliant, and cooperated with follow-up visits.

(B) The provider must fulfill the following conditions:

1. Age greater than or equal to 12 years;
2. HLA mating types are at least hemi-compatible;
3. Adequate venous access is available for peripheral blood leukocyte isolation;
4. Voluntary written informed consent.

Exclusion criteria

(A) Subjects who meet any of the following criteria are not eligible for enrollment in this study

1. Patients who have used CAR-T cell therapy or any other therapeutic product such as gene transduction within 3 months of signing the informed consent, except for those with undetectable CAR-T or CAR-T below the lower limit of detection; or patients who have participated in an interventional clinical study of an antitumor drug within 4 weeks prior to signing the informed consent;
2. Individuals with a history of any of the following cardiovascular diseases within 6 months prior to screening: (1) congestive heart failure (New York Heart Association [NYHA] class ≥III), myocardial infarction, unstable angina, congenital long QT syndrome, left anterior hemiblock (bifascicular block), coronary angioplasty, stenting, coronary/peripheral artery bypass grafting, cerebrovascular accident ( CVA), transient ischemic attack, or pulmonary embolism, allowing for asymptomatic right bundle branch block; (2) severe cardiac arrhythmias requiring treatment (e.g., sustained ventricular tachycardia, ventricular fibrillation, tip-twist ventricular tachycardia, etc.); and (3) suffering from uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), a history of hypertensive crisis, or hypertensive encephalopathy;
3. Hepatitis B surface antigen (HBsAg) positive, Hepatitis B core antibody (HBcAb) positive subjects with peripheral blood HBV DNA copy number higher than the limit of detection, Hepatitis C virus (HCV) antibody positive subjects with HCV RNA copy number higher than the limit of detection, and Syphilis spirochete antibody test positive subjects;
4. Patients with known systemic lupus erythematosus, comorbid active or uncontrolled autoimmune diseases (e.g., Crohns disease, rheumatoid arthritis, autoimmune hemolytic anemia, etc.), and primary or secondary immunodeficiencies (e.g., HIV infection or severe infectious diseases, etc.);
5. Pre-existing or concurrent other untreated malignancies of indolent control affecting the subject's long-term survival, except cured carcinoma in situ of the uterine cervix, non-invasive basal cell or squamous cell skin cancers, or other malignancies that have been radically treated with localized prostate cancer, or ductal carcinoma in situ after radical surgery, and that have remained free of recurrence for at least 5 years;
6. Patients with current or previous history of CNS disorders such as seizures, stroke, severe brain injury aphasia, paralysis, dementia, Parkinson's disease, psychiatric disorders;
7. Those with active central nervous system leukemia (CNSL) present at screening;
8. History of solid organ transplantation or hematopoietic stem cell transplantation (HSCT) within 6 months prior to screening;
9. Those with acute or chronic graft-versus-host disease (GVHD) at screening;
10. Use of patients who have had any of the following medications or treatments performed within the designated time period prior to single-take:

    * Have used any immunosuppressant within 2 weeks prior to single harvesting;
    * Received any chemotherapy or small molecule targeted therapy within 2 weeks or 3 half-lives (whichever is shorter) prior to monoacquisition;
    * Received any large molecule therapy such as monoclonal antibody, antibody coupled drug (ADC), or doublet within 4 weeks or 3 half-lives (whichever is shorter) prior to monoacquisition;
11. People with mental illness, or a history of substance abuse;
12. Pregnant or lactating subjects;
13. Other factors that, in the opinion of the investigator, make enrollment inappropriate or affect the subject's participation in or completion of the study.

(B) Donor exclusion criteria

Any of the following points are used as provider/third party exclusion criteria:

1. A history of mental disorder that may interfere with compliance with the program or prevent signing the informed consent form;
2. History of uncontrollable high blood pressure with medication, stroke or severe heart disease;
3. There is anemia or thrombocytopenia;
4. HBsAg-positive, or HBcAb-positive and peripheral blood HBV DNA-positive; HCV-antibody-positive individuals and HCV RNA-positive; syphilis spirochete antibody-positive; HIV antibody-positive;
5. Presence or suspicion of uncontrolled fungal, bacterial, viral or other infections;
6. Pregnancy;
7. Any other circumstances that the investigator deems inappropriate as a donor/third party.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability | 12 months
  Subjects are observed for dose-limiting toxicity(DLT) after LILRB4 STAR-T cells infusion, with the recording of adverse events(AE) and serious adverse events(SAE), with a focus on cytokine release syndrome(CRS) and immune cell-associated neurotoxicity(ICANS).All of the AE ratings were assessed according to the CTCAE.

SECONDARY OUTCOMES:
Describe preliminaryefficacy of LILRB4 STAR-T cells | 12 months
  Duration of Response (DOR)
Rate of morphologic complete remission (CR) | 12 months
  Bone marrow blasts < 5%, absence of blasts with Auer rods, absence ofextramedullary disease; absolute neutrophil count >1.0G/L(1000/uL); plateletcount >100 xG/L(100.000/uL);independence of red cell transfusions.
Describe preliminaryefficacy of LILRB4 STAR-T cells | 12 months
  Overall Survival (OS)
Describe preliminaryefficacy of LILRB4 STAR-T cells | 12 months
  Overall response rate
Describe preliminaryefficacy of LILRB4 STAR-T cells | 12 months
  Recurrence free survival（RFS）
Describe preliminaryefficacy of LILRB4 STAR-T cells | 12 months
  Event-free lifetime（EFS）

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Zhao, Principal Investigator — PEKING UNICERSITY PEOPLE'S HOSPITAL
Locations (2):
- China (2):
  - Peking Unicersity People'S Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No